CLINICAL TRIAL: NCT04804033
Title: A Phase 2/3 Randomized, Double-Blind, Placebo- Controlled Study to Evaluate the Efficacy and Safety of Oral Zavegepant in Migraine Prevention
Brief Title: A Study to Evaluate the Efficacy and Safety of Oral Zavegepant in Migraine Prevention
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Strategic decision to discontinue the study based on adjusted clinical development plan. This decision is not based on any safety concerns.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: BHV3500-302; C5301006 (Other: Alias Study Number)
Record Dates: First submitted 2021-03-05; First posted 2021-03-18 (Actual); Results first posted 2025-03-27 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Migraine
Keywords: Migraine Prevention; Phonophobia; Photophobia; Nausea
MeSH Terms: conditions — Migraine Disorders; Hyperacusis; Photophobia; Nausea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- BHV-3500 200mg (Active Comparator): Zavegepant 200mg oral soft gel capsule.
  Interventions: Drug: BHV-3500 (zavegepant)
- Placebo 200mg (Placebo Comparator): Matching placebo 200mg oral soft gel capsule.
  Interventions: Drug: Placebo
- BHV-3500 100mg (Active Comparator): Zavegepant 100mg oral soft gel capsule.
  Interventions: Drug: BHV-3500 (zavegepant)
- Placebo 100mg (Placebo Comparator): Matching placebo 100mg oral soft gel capsule.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BHV-3500 (zavegepant) — BHV-3500 (zavegepant) softgel capsule.
  Arms: BHV-3500 100mg; BHV-3500 200mg
Drug: Placebo — Matching placebo softgel capsule.
  Arms: Placebo 100mg; Placebo 200mg

SUMMARY:
The purpose of this is study is to compare the efficacy of BHV-3500 (zavegepant) to placebo as a preventive treatment for migraine, as measured by the reduction in the number of migraine days per month.

ELIGIBILITY:
Inclusion Criteria:

Subject has at least 1 year history of migraine (with or without aura) consistent with a diagnosis according to the International Classification of

Headache Disorders, 3rd Edition, including the following:

1. Age of onset of migraines prior to 50 years of age
2. Migraine attacks, on average, lasting 4 - 72 hours if untreated
3. Per subject report, at least 15 headache days per month, at lest 8 migraine days per month, and at least 1 headache-free day per month within the last 3 months prior to the Screening Visit
4. Eight or more migraine days during the Observation Period
5. 15 or more headache days during the Observation Period
6. One or more non-headache days during the Observation Period
7. Ability to distinguish migraine attacks from tension/cluster headaches
8. Subjects on prophylactic migraine medication are permitted to remain on 1 medication with possible migraine-prophylactic effects if the dose has been stable for at least 3 months prior to the Screening Visit, and the dose is not expected to change during the course of the study.

Exclusion Criteria:

1. Subject with a history of HIV disease
2. Subject history with current evidence of uncontrolled, unstable or recently diagnosed cardiovascular disease, such as ischemic heart disease, coronary artery vasospasm, and cerebral ischemia. Subjects with Myocardial Infarction (MI), Acute Coronary Syndrome (ACS), Percutaneous Coronary Intervention (PCI), cardiac surgery, stroke or transient ischemic attack (TIA) during the 6 months prior to screening
3. Uncontrolled hypertension (high blood pressure), or uncontrolled diabetes (however subjects can be included who have stable hypertension and/or diabetes for at least 3 months prior to screening).
4. Subjects with major depressive episode or anxiety disorder which require more than 1 daily medication for each disorder or subjects with a major depressive episode within the last 12 months. Medications to treat major depressive disorder or an anxiety disorder must have been at a stable dose for at least 3 months prior to the Screening Visit.
5. Subjects with active chronic pain syndromes, other pain syndromes (including trigeminal neuralgia), psychiatric conditions, dementia, or significant neurological disorders (other than migraine) that, in the Investigator's opinion interfere with study assessments of safety or efficacy.
6. Subject has a history of gastric, or small intestinal surgery (including Gastric Bypass, Gastric Banding, Gastric Sleeve, Gastric Balloon, etc.), or has disease or condition (e.g. chronic pancreatitis, ulcerative colitis, etc.) that causes malabsorption.
7. Body mass index > 33 kg/m2
8. History of gallstones or cholecystectomy.
9. The subject has a history or current evidence of any unstable medical conditions (e.g., history of congenital heart disease or arrhythmia, known or suspected infection, hepatitis B or C, or cancer) that, in the investigator's opinion, would expose them to undue risk of a significant adverse event (AE) or interfere with assessments of safety or efficacy during the course of the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1753 (Actual)
Dates: Start 2021-03-26 (Actual); Primary Completion 2024-03-21 (Actual); Study Completion 2024-03-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (113):
- United States (113):
  - Xenoscience, Inc, Phoenix, Arizona
  - Tucson Neuroscience Research, Tucson, Arizona
  - Hope Clinical Research, Canoga Park, California
  - Axiom Research, Llc, Colton, California
  - Wr-Pri, Llc, Encino, California
  - eStudySite, La Mesa, California
  - Synergy San Diego, Lemon Grove, California
  - Collaborative Neuroscience Research, LLC., Long Beach, California
  - Clinical Research Institute, Los Angeles, California
  - Wr-Pri, Llc, Newport Beach, California
  - Artemis Institute for Clinical Research, San Diego, California
  - California Neuroscience Research Medical Group, inc., Sherman Oaks, California
  - CMR of Greater New Haven, LLC, Hamden, Connecticut
  - Ki Health Partners, LLc, dba New England Institute for Clinical Research, Stamford, Connecticut
  - Chase Medical Research, LLC, Waterbury, Connecticut
  - Neurology Offices of South Florida, Boca Raton, Florida
  - Accel Research Sites Network - Edgewater Clinical Research Unit, Edgewater, Florida
  - Complete Health Research, Edgewater, Florida
  - Sarkis Clinical Trials, Gainesville, Florida
  - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - Multi-Specialty Research Associates, Inc., Lake City, Florida
  - AppleMed Research Group, LLC, Miami, Florida
  - Brainstorm Research, Miami, Florida
  - The Neurology Research Group, Miami, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - Complete Health Research, Ormond Beach, Florida
  - Ideal Clinical Research, Pembroke Pines, Florida
  - Clinical Research Center of Florida, Pompano Beach, Florida
  - Clin-Med Research & Development LLC, South Miami, Florida
  - Accel Research Sites Network - St. Petersburg Clinical Research Unit, St. Petersburg, Florida
  - ForCare Clinical Research, Tampa, Florida
  - JSV Clinical Research Study Inc, Tampa, Florida
  - CenExel iResearch, LLC, Decatur, Georgia
  - iResearch Atlanta LLC, Decatur, Georgia
  - Cedar Crosse Research Center, Chicago, Illinois
  - Clinical Investigation Specialists, Inc., Gurnee, Illinois
  - Clinical Investigation Specialists, Inc, Gurnee, Illinois
  - MediSphere Medical Research Center, LLC., Evansville, Indiana
  - MediSphere Medical Research Center, LLC, Evansville, Indiana
  - Meridian Clinical Research, LLC, Sioux City, Iowa
  - Alliance for Multispecialty Reseach, LLC, El Dorado, Kansas
  - Alliance for Multispecialty Research, LLC, Newton, Kansas
  - Collevtive Medical Research, Overland Park, Kansas
  - Kansas Institute of Research, Overland Park, Kansas
  - The Research Group of Lexington, Llc., Lexington, Kentucky
  - The Research Group of Lexington, Llc, Lexington, Kentucky
  - L-MARC Research Center, Louisville, Kentucky
  - Crescent City Headache and Neurology Center, Chalmette, Louisiana
  - Alliance for Multispecialty Research, LLC., New Orleans, Louisiana
  - DelRicht Research, New Orleans, Louisiana
  - Boston Clinical Trials, Boston, Massachusetts
  - Neurology Center of New England P.C., Foxborough, Massachusetts
  - Community Clinical Research Network Inc, Marlborough, Massachusetts
  - MedVadis Research Corporation, Waltham, Massachusetts
  - Michigan Head Pain & Neurological Institute, Ann Arbor, Michigan
  - Romedica LLC, Rochester, Michigan
  - StudyMetrix Research, City of Saint Peters, Missouri
  - Alliance for Multispecialty Reseach, LLC, Kansas City, Missouri
  - Clinvest Research, LLC, Springfield, Missouri
  - Meridian Clinical Research, LLC, Norfolk, Nebraska
  - Excel Clinical research, Las Vegas, Nevada
  - Wr-Crcn, Llc, Las Vegas, Nevada
  - Albuquerque Clinical Trials, Inc., Albuquerque, New Mexico
  - Dent Neurosciences Research Center, Inc., Amherst, New York
  - Central New York Clinical Research, Manlius, New York
  - New York Neurology Associates, New York, New York
  - Fieve Clinical Research, Inc, New York, New York
  - North Suffolk Neurology, PC, Port Jefferson Station, New York
  - Montefiore Medical Center, The Bronx, New York
  - Upstate Clinical Research Associates, LLC, Williamsville, New York
  - Headache Wellness Center, Greensboro, North Carolina
  - Accellacare, Raleigh, North Carolina
  - M3 Wake Research, Inc., Raleigh, North Carolina
  - Carolina Research Center, Inc., Shelby, North Carolina
  - Accellacare, Wilmington, North Carolina
  - CTI Clinical Research Center, Cincinnati, Ohio
  - WellNow Urgent Care and Research, Cincinnati, Ohio
  - Wellnow Urgent Care, Cincinnati, Ohio
  - Hometown Urgent Care and Research, Columbus, Ohio
  - Wellnow Urgent Care and Research, Columbus, Ohio
  - Hometown Urgent Care and Research, Dayton, Ohio
  - WellNow Urgent Care and Research, Dayton, Ohio
  - Neuro-Behavioral Clinical Research, Inc., North Canton, Ohio
  - WellNow Urgent Care and Research, Troy, Ohio
  - Hightower Clinical, Oklahoma City, Oklahoma
  - Summit Headlands LLC, dba Summit Research, Portland, Oregon
  - Clinical Research Philadelphia, LLC, Philadelphia, Pennsylvania
  - Preferred Primary Care Physicians, Inc., Pittsburgh, Pennsylvania
  - Preferred Primary Care Physicians, Uniontown, Pennsylvania
  - Reading Hospital Clinical Trials Office, West Reading, Pennsylvania
  - Tower Health Medical Group - Neurology, West Reading, Pennsylvania
  - Coastal Carolina Research Center, North Charleston, South Carolina
  - Accellacare (Administrative Only), Bristol, Tennessee
  - Internal Medicine and Pediatric Associates of Bristol, PC, Bristol, Tennessee
  - WR-ClinSearch, LLC, Chattanooga, Tennessee
  - KCA Neurology, PLLC, Franklin, Tennessee
  - Clinical Neuroscience Solutions, Inc., Memphis, Tennessee
  - FutureSearch Trials of Neurology, Austin, Texas
  - FutureSearch Trials of Dallas, LP, Dallas, Texas
  - North Texas Institute of Neurology and Headache - NextStage Clinical Research, Frisco, Texas
  - North Texas Institute of Neurology and Headache, Frisco, Texas
  - Texas Center for Drug Development, Inc., Houston, Texas
  - Red Star Research. LLC, Lake Jackson, Texas
  - FMC Science, Lampasas, Texas
  - Radiance Clinical Research, Lampasas, Texas
  - DM Clinical Research, Tomball, Texas
  - Wasatch Clinical Research , LLC(Administrative Location), Salt Lake City, Utah
  - Charlottesville Medical Research Center, LLC, Charlottesville, Virginia
  - Health Research of Hampton Roads, Inc., Newport News, Virginia
  - Meridian Clinical Research, LLC, Norfolk, Virginia
  - Northwest Clinical Research Center, Bellevue, Washington
  - Seattle Clinical Research Center, Seattle, Washington
  - Seattle Women's: Health, Research, Gynecology, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=BHV3500-302

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study enrolled 1753 participants, out of which 1219 were not randomized. Only 534 participants were randomized in a 12-week double-blind treatment (DBT) phase. A total of 298 eligible participants then entered in a 52-week open-label extension (OLE) phase. Participants had a follow-up of 8 weeks after discontinuation or completion of treatment in DBT (if not entered OLE) or OLE phase.
Groups:
- Zavegepant 100 mg (OLE/DBT): Participants were randomized to receive Zavegepant 100 milligrams (mg) orally as soft gelatin capsules (25 mg *4 capsules) daily for 12 weeks in DBT phase. Eligible participants continued to receive Zavegepant in similar manner for another 52 weeks in OLE phase.
- Zavegepant 200 mg (OLE/DBT): Participants were randomized to receive Zavegepant 200 mg orally as soft gelatin capsules (25 mg *8 capsules) daily for 12 weeks in DBT phase. Eligible participants continued to receive Zavegepant in similar manner for another 52 weeks in OLE phase.
- Placebo (DBT)/ Zavegepant 100 mg (OLE): Participants were randomized to receive placebo matched to Zavegepant 100 mg daily for 12 weeks in DBT phase. Eligible participants received Zavegepant 100 mg orally as soft gelatin capsules (25 mg *4 capsules) daily for 52 weeks in OLE phase.
- Placebo (DBT)/ Zavegepant 200 mg (OLE): Participants were randomized to receive placebo matched to Zavegepant 200 mg daily for 12 weeks in DBT phase. Eligible participants received Zavegepant 200 mg orally as soft gelatin capsules (25 mg *8 capsules) daily for 52 weeks in OLE phase.
Period: Period 1: DBT Phase
Arm/Group | Zavegepant 100 mg (OLE/DBT) | Zavegepant 200 mg (OLE/DBT) | Placebo (DBT)/ Zavegepant 100 mg (OLE) | Placebo (DBT)/ Zavegepant 200 mg (OLE)
Started | 178 | 180 | 88 | 88
Treated | 173 | 175 | 86 | 88
Completed | 144 | 134 | 69 | 64
Not Completed | 34 | 46 | 19 | 24
Not completed — Adverse Event | 1 | 5 | 3 | 4
Not completed — Death | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 3 | 7 | 1 | 3
Not completed — Non-compliance | 1 | 0 | 1 | 2
Not completed — Other | 0 | 1 | 0 | 0
Not completed — Pregnancy | 2 | 0 | 0 | 0
Not completed — Study terminated by sponsor | 15 | 16 | 5 | 9
Not completed — Withdrawal by Subject | 6 | 12 | 7 | 6
Not completed — Randomized but not treated | 5 | 5 | 2 | 0
Period: Period 2: OLE Phase
Arm/Group | Zavegepant 100 mg (OLE/DBT) | Zavegepant 200 mg (OLE/DBT) | Placebo (DBT)/ Zavegepant 100 mg (OLE) | Placebo (DBT)/ Zavegepant 200 mg (OLE)
Started | 105 (Eligible participants who completed DBT phase and entered the OLE phase.) | 94 (Eligible participants who completed DBT phase and entered the OLE phase.) | 50 (Eligible participants who completed DBT phase and entered the OLE phase.) | 49 (Eligible participants who completed DBT phase and entered the OLE phase.)
Treated | 105 | 94 | 50 | 49
Completed | 34 | 34 | 22 | 17
Not Completed | 71 | 60 | 28 | 32
Not completed — Adverse Event | 3 | 4 | 2 | 0
Not completed — Lost to Follow-up | 8 | 4 | 3 | 4
Not completed — Non-compliance | 2 | 2 | 0 | 1
Not completed — Other | 0 | 2 | 0 | 0
Not completed — Physician Decision | 1 | 1 | 0 | 0
Not completed — Pregnancy | 0 | 0 | 2 | 0
Not completed — Study terminated by sponsor | 41 | 37 | 17 | 19
Not completed — Withdrawal by Subject | 16 | 8 | 3 | 7
Not completed — Not reported | 0 | 2 | 0 | 0
Not completed — Failure to meet continuation criteria | 0 | 0 | 1 | 1
Period: Period 3: Follow-up Phase
Arm/Group | Zavegepant 100 mg (OLE/DBT) | Zavegepant 200 mg (OLE/DBT) | Placebo (DBT)/ Zavegepant 100 mg (OLE) | Placebo (DBT)/ Zavegepant 200 mg (OLE)
Started | 154 (Eligible participants who entered follow-up phase either directly from DBT phase or after OLE phase.) | 162 (Eligible participants who entered follow-up phase either directly from DBT phase or after OLE phase.) | 47 (Eligible participants who entered follow-up phase either directly from DBT phase or after OLE phase.) | 48 (Eligible participants who entered follow-up phase either directly from DBT phase or after OLE phase.)
Completed | 124 | 131 | 41 | 38
Not Completed | 30 | 31 | 6 | 10
Not completed — Lost to Follow-up | 5 | 9 | 0 | 1
Not completed — Other | 0 | 1 | 2 | 1
Not completed — Withdrawal by Subject | 7 | 6 | 3 | 4
Not completed — Not reported | 18 | 15 | 1 | 4

BASELINE CHARACTERISTICS:
Population: DBT safety analysis set included participants in the safety analysis set who took greater than or equal to (>=) 1 dose of DB study drug (zavegepant or placebo), i.e., nonmissing DB study drug start date.
Groups:
- Zavegepant 100 mg (DBT): Participants were randomized to receive Zavegepant 100 milligrams (mg) orally as soft gelatin capsules (25 mg *4 capsules) daily for 12 weeks in DBT phase.
- Zavegepant 200 mg (DBT): Participants were randomized to receive Zavegepant 200 mg orally as soft gelatin capsules (25 mg *8 capsules) daily for 12 weeks in DBT phase.
- Placebo (DBT) Matched to Zavegepant 100 mg: Participants were randomized to receive placebo matched to Zavegepant 100 mg daily for 12 weeks in DBT phase.
- Placebo (DBT) Matched to Zavegepant 200 mg: Participants were randomized to receive placebo matched to Zavegepant 200 mg daily for 12 weeks in DBT phase.
- Total: Total of all reporting groups
Arm/Group | Zavegepant 100 mg (DBT) | Zavegepant 200 mg (DBT) | Placebo (DBT) Matched to Zavegepant 100 mg | Placebo (DBT) Matched to Zavegepant 200 mg | Total
Number analyzed (Participants) | 173 | 175 | 86 | 88 | 522
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.7 (12.85) | 43.2 (13.30) | 41.7 (13.15) | 41.5 (13.14) | 42.2 (13.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 127 | 144 | 72 | 70 | 413
  Male | 46 | 31 | 14 | 18 | 109
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 48 | 47 | 26 | 27 | 148
  Not Hispanic or Latino | 125 | 128 | 60 | 61 | 374
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 1
  Asian | 4 | 2 | 3 | 5 | 14
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 0 | 1 | 3
  Black or African American | 35 | 35 | 16 | 17 | 103
  White | 130 | 132 | 66 | 63 | 391
  More than one race | 4 | 4 | 1 | 0 | 9
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Observation Phase (OP) in the Number of Migraine Days Per Month Over Entire DBT Phase (Weeks 1 to 12)
Description: A migraine day was defined as any calendar day in which participant experienced a qualified migraine headache (onset, continuation or recurrence of migraine headache). A qualified migraine headache was defined as migraine with or without aura, lasting for greater than or equal to (>=) 30 minutes, and met at least one of the following criteria (A and/or B): A. >=2 of the following pain features: a. Unilateral location, b. Pulsating quality (throbbing), c. Moderate or severe pain intensity, d. Aggravation by or causing avoidance of routine physical activity (e.g. walking or climbing stairs) B. >= 1 of following associated symptoms: a. Nausea and/or vomiting b. Photophobia and phonophobia. The number of migraine days per month were prorated to 28 days and derived as follows: 28*(total number of migraine days through Month 3[Weeks 1 to 12] in on-DBT efficacy analysis period)/ (total number of eDiary efficacy data days through Month 3[Weeks 1 to 12] in the on-DBT efficacy analysis period).
Time Frame: Observation Phase: 28 days prior to randomization and baseline; Entire DBT Phase: 12 weeks (Week 1 through 12)
Population: Migraine analysis set included participants in the DBT efficacy analysis set with >= 14 days of e-diary efficacy data in both the observation phase and >= 1 month (4-week interval) in the DBT phase. DBT efficacy analysis set: participants who were enrolled and randomized only once and took >=1 dose of DB study drug (zavegepant or placebo). Results were summarized by treatment group and the 2 matching placebo groups were pooled as pre-specified in protocol/ statistical analysis plan (SAP).
Measure: Least Squares Mean (97.5% Confidence Interval); unit: Migraine Days per Month
Groups:
- Placebo Pooled (DBT): Participants were randomized to receive placebo matched to Zavegepant 100 mg or 200 mg daily for 12 weeks in DBT phase.
Arm/Group | Zavegepant 100 mg (DBT) | Zavegepant 200 mg (DBT) | Placebo Pooled (DBT)
Number analyzed (Participants) | 164 | 163 | 165
Migraine Days per Month | -7.0 [-8.10 to -5.92] | -6.3 [-7.45 to -5.10] | -5.6 [-6.80 to -4.37]
Statistical Analysis 1: Comparison: Zavegepant 100 mg (DBT) vs Placebo Pooled (DBT); Test type: Other; Difference in least square mean (LSM) = -1.4, 97.5% CI 2-sided [-2.72 to -0.12] — Linear mixed effects model with repeated measures with number of total migraine days per month in the OP as covariate, treatment group, randomization stratum, month, month-by treatment group interaction as fixed effects using migraine analysis set
Statistical Analysis 2: Comparison: Zavegepant 200 mg (DBT) vs Placebo Pooled (DBT); Test type: Other; Difference in LSM = -0.7, 97.5% CI 2-sided [-2.07 to 0.69] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Percentage of Participants With >= 50 % Reduction in Number of Moderate to Severe Migraine Days Per Month Over Entire DBT Phase (Weeks 1 to 12)
Description: A migraine day was defined as any calendar day in which participant experienced a qualified migraine headache (onset, continuation or recurrence of the migraine headache). A qualified migraine headache was defined as migraine with or without aura, lasting for greater than or equal to (>=) 30 minutes, and met at least one of following criteria (A and/or B): A. >=2 of following pain features: a. Unilateral location, b. Pulsating quality (throbbing), c. Moderate or severe pain intensity, d. Aggravation by or causing avoidance of routine physical activity (e.g. walking or climbing stairs) B. >= 1 of the following associated symptoms: a. Nausea and/or vomiting b. Photophobia and phonophobia. The number of migraine days per month were prorated to 28 days and derived as follows: 28*(total number of migraine days through Month 3[Weeks 1 to 12] in the on-DBT efficacy analysis period)/ (total number of eDiary efficacy data days through Month 3[Weeks 1 to 12] in on-DBT efficacy analysis period).
Time Frame: Entire DBT Phase: 12 weeks (Week 1 through 12)
Population: Migraine analysis set included participants in the DBT efficacy analysis set with >= 14 days of e-diary efficacy data in both the observation phase and >= 1 month (4-week interval) in the DBT phase. DBT efficacy analysis set: participants who were enrolled and randomized only once and took >=1 dose of DB study drug (zavegepant or placebo). Results were summarized by treatment group and the 2 matching placebo groups were pooled as pre-specified in protocol/ SAP.
Measure: Number (97.5% Confidence Interval); unit: Percentage of participants
Arm/Group | Zavegepant 100 mg (DBT) | Zavegepant 200 mg (DBT) | Placebo Pooled (DBT)
Number analyzed (Participants) | 164 | 163 | 165
Percentage of participants | 56.1 [47.7 to 65.1] | 46.6 [37.8 to 55.4] | 40.0 [31.4 to 48.5]
Statistical Analysis 1: Comparison: Zavegepant 100 mg (DBT) vs Placebo Pooled (DBT); Test type: Other; Difference in percentage = 16.6, 97.5% CI 2-sided [4.4 to 28.8] — Stratified by randomization stratum using Mantel-Haenszel risk estimation
Statistical Analysis 2: Comparison: Zavegepant 200 mg (DBT) vs Placebo Pooled (DBT); Test type: Other; Difference in percentage = 6.6, 97.5% CI 2-sided [-5.6 to 18.9] — Stratified by randomization stratum using Mantel-Haenszel risk estimation

3. Secondary Outcome: Mean Change From Observation Phase in the Number of Migraine Days Per Month in the Last 4 Weeks (Weeks 9 to 12) of DBT Phase
Description: A migraine day was defined as any calendar day in which the participant experienced a qualified migraine headache (onset, continuation or recurrence of the migraine headache). A qualified migraine headache was defined as a migraine with or without aura, lasting for greater than or equal to (>=) 30 minutes, and met at least one of the following criteria (A and/or B): A.>=2 of the following pain features: a. Unilateral location, b. Pulsating quality (throbbing), c. Moderate or severe pain intensity, d. Aggravation by or causing avoidance of routine physical activity (e.g. walking or climbing stairs) B. >= 1 of the following associated symptoms: a. Nausea and/or vomiting b. Photophobia and phonophobia. The number of migraine days per month were prorated to 28 days and derived for month (i.e., 4-week interval) in on-DBT efficacy analysis period as follows: 28* (total number of migraine days in the month[Week 9 to 12])/(total number of eDiary efficacy data days in the month[Week 9 to 12]).
Time Frame: Observation Phase: 28 days prior to randomization and baseline; DBT Phase: last 4 weeks (Week 9 through 12)
Population: Migraine analysis set analyzed. Here, "Overall Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure. Results were summarized by treatment group and the 2 matching placebo groups were pooled as pre-specified in protocol/ SAP.
Measure: Least Squares Mean (97.5% Confidence Interval); unit: Migraine Days per Month
Groups:
- Placebo Pooled: Participants received 100 mg and 200 mg daily dose of 4 oral soft gel capsules for up to 52-weeks.
Arm/Group | Zavegepant 100 mg (DBT) | Zavegepant 200 mg (DBT) | Placebo Pooled
Number analyzed (Participants) | 137 | 123 | 126
Migraine Days per Month | -7.8 [-9.11 to -6.59] | -7.2 [-8.56 to -5.83] | -6.8 [-8.22 to -5.38]
Statistical Analysis 1: Comparison: Zavegepant 100 mg (DBT) vs Placebo Pooled; Test type: Other; Difference in LSM = -1, 97.5% CI 2-sided [-2.68 to 0.58] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Zavegepant 200 mg (DBT) vs Placebo Pooled; Test type: Other; Difference in LSM = -0.4, 97.5% CI 2-sided [-2.10 to 1.31] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Mean Change From Observation Phase in the Number of Migraine Days Per Month in the First 4 Weeks (Weeks 1 to 4) of DBT Phase
Description: A migraine day was defined as any calendar day in which participant experienced a qualified migraine headache (onset, continuation or recurrence of the migraine headache). A qualified migraine headache was defined as a migraine with or without aura, lasting for greater than or equal to (>=) 30 minutes, and met at least one of the following criteria (A and/or B): A. >=2 of the following pain features: a. Unilateral location, b. Pulsating quality (throbbing), c. Moderate or severe pain intensity, d. Aggravation by or causing avoidance of routine physical activity (e.g. walking or climbing stairs) B. >= 1 of the following associated symptoms: a. Nausea and/or vomiting b. Photophobia and phonophobia. The number of migraine days per month were prorated to 28 days and derived for month (i.e., 4-week interval) in the on-DBT efficacy analysis period as follows: 28* (total number of migraine days in the month[Week 1 to 4])/ (total number of eDiary efficacy data days in the month[Week 1 to 4]).
Time Frame: Observation Phase: 28 days prior to randomization and baseline; DBT Phase: first 4 weeks (Week 1 through 4)
Population: Migraine analysis set analyzed. Results were summarized by treatment group and the 2 matching placebo groups were pooled as pre-specified in protocol/ SAP. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Least Squares Mean (97.5% Confidence Interval); unit: Migraine Days per Month
Arm/Group | Zavegepant 100 mg (DBT) | Zavegepant 200 mg (DBT) | Placebo Pooled (DBT)
Number analyzed (Participants) | 162 | 161 | 164
Migraine Days per Month | -5.7 [-6.89 to -4.51] | -5.1 [-6.26 to -3.87] | -3.9 [-5.10 to -2.72]
Statistical Analysis 1: Comparison: Zavegepant 100 mg (DBT) vs Placebo Pooled (DBT); Test type: Other; Difference in LSM = -1.8, 97.5% CI 2-sided [-3.16 to -0.42] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Zavegepant 200 mg (DBT) vs Placebo Pooled (DBT); Test type: Other; Difference in LSM = -1.2, 97.5% CI 2-sided [-2.53 to 0.22] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Mean Number of Acute Migraine -Specific Medication Days Per Month Over Entire DBT Phase (Weeks 1 to 12)
Description: Acute migraine (AM)-specific medication day was defined as any calendar day on which the participant took an acute migraine-specific medication during aura or to treat a headache. Acute migraine-specific medications were triptans and ergotamine. The number of acute migraine-specific medication days per month were prorated to 28 days and derived as follows: 28 * (total number of acute migraine-specific medication days through Month 3 [Week 1 to 12] in the on-DBT efficacy analysis period)/ (total number of eDiary efficacy data days through Month 3 [Week 1 to 12] in the on-DBT efficacy analysis period).
Time Frame: Entire DBT Phase: 12 weeks (Week 1 through 12)
Population: as for outcome 2
Measure: Least Squares Mean (97.5% Confidence Interval); unit: AM-specific Medication Days per Month
Arm/Group | Zavegepant 100 mg (DBT) | Zavegepant 200 mg (DBT) | Placebo Pooled (DBT)
Number analyzed (Participants) | 164 | 163 | 165
AM-specific Medication Days per Month | 2.4 [1.43 to 3.43] | 3.0 [1.91 to 4.17] | 3.2 [1.94 to 4.46]
Statistical Analysis 1: Comparison: Zavegepant 100 mg (DBT) vs Placebo Pooled (DBT); Test type: Other; Difference in LSM = -0.8, 97.5% CI 2-sided [-1.59 to 0.05] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Zavegepant 200 mg (DBT) vs Placebo Pooled (DBT); Test type: Other; Difference in LSM = -0.2, 97.5% CI 2-sided [-1.06 to 0.74] — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Mean Change From Baseline in the Migraine-specific Quality of Life Questionnaire (MSQ) v 2.1 Restrictive Role Function Domain Score at Week 12
Description: MSQ v 2.1 is 14-item questionnaire that assessed impact of treatment on participant-reported quality of life across 3 domains: role function-restrictive, preventive, and emotional function. Restrictive role function domain consists of 7 items that describe how migraine limits one's daily social, work-related activities. Participants respond to items using a 6-point scale ranging from 1 (none of the time) to 6 (all of the time), which are assigned scores of 1 to 6, respectively. Response from each item of restrictive role function domain were added providing a possible raw score range of 7 (no impairment) to 42 (maximum impairment). Raw score range of restrictive role function domain was then transformed to a 0 (no impairment) to 100 (maximum impairment), higher scores = higher impairment.
Time Frame: DBT Phase: Baseline (before dose on Day 1), Week 12
Population: DBT efficacy analysis set included participants in the full analysis set who were randomized only once and took >= 1 dose of DB study drug (zavegepant or placebo). Here, " Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure. Results were summarized by treatment group and the 2 matching placebo groups were pooled as pre-specified in protocol/ SAP.
Measure: Least Squares Mean (97.5% Confidence Interval); unit: Scores on a scale
Arm/Group | Zavegepant 100 mg (DBT) | Zavegepant 200 mg (DBT) | Placebo Pooled (DBT)
Number analyzed (Participants) | 143 | 125 | 136
Scores on a scale | 24.5 [19.10 to 29.83] | 20.6 [14.63 to 26.61] | 20.5 [14.92 to 26.12]
Statistical Analysis 1: Comparison: Zavegepant 100 mg (DBT) vs Placebo Pooled (DBT); Test type: Other; Difference in LSM = 3.9, 97.5% CI 2-sided [-1.50 to 9.39] — Linear regression model had the following variables: Week 12 change from baseline in domain score as the dependent variable; baseline domain score as a covariate; treatment group and randomization stratum as fixed effects
Statistical Analysis 2: Comparison: Zavegepant 200 mg (DBT) vs Placebo Pooled (DBT); Test type: Other; Difference in LSM = 0.1, 97.5% CI 2-sided [-5.66 to 5.86] — [estimate comment as in outcome 6, analysis 1]

7. Secondary Outcome: Mean Change From Baseline in the Migraine Disability Assessment (MIDAS) Total Score at Week 12
Description: MIDAS is a retrospective, participant-reported, 5-item questionnaire that measured headache related disability as lost days due to headache from paid work or school, household work and non-work activities over past 3-months. The total score is calculated as the sum of item scores to all 5 questions on a scale of 0 (no disability) to 90 (maximum disability) resulting into overall possible MIDAS total score (range from 0 (no disability) to 450 (maximum disability). Higher scores = more severe disability.
Time Frame: DBT Phase: Baseline (before dose on Day 1), Week 12
Population: as for outcome 6
Measure: Least Squares Mean (97.5% Confidence Interval); unit: Scores on a scale
Arm/Group | Zavegepant 100 mg (DBT) | Zavegepant 200 mg (DBT) | Placebo Pooled (DBT)
Number analyzed (Participants) | 143 | 125 | 135
Scores on a scale | -26.8 [-35.81 to -17.79] | -27.1 [-36.62 to -17.61] | -17.9 [-31.36 to -4.34]
Statistical Analysis 1: Comparison: Zavegepant 100 mg (DBT) vs Placebo Pooled (DBT); Test type: Other; Difference in LSM = -9, 97.5% CI 2-sided [-18.10 to 0.19] — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 2: Comparison: Zavegepant 200 mg (DBT) vs Placebo Pooled (DBT); Test type: Other; Difference in LSM = -9.3, 97.5% CI 2-sided [-18.95 to 0.41] — [estimate comment as in outcome 6, analysis 1]

8. Secondary Outcome: Number of Participants With Moderate or Severe Adverse Events (AEs): DBT Phase
Description: AEs: new untoward medical occurrence or worsening of a pre-existing medical condition in participant or clinical investigation participant administered investigational product that does not necessarily have a causal relationship with treatment. AEs included both SAEs and all non-SAEs. Severity: Moderate=Alleviated with additional specific therapeutic intervention, interfered with activities of daily living, causing discomfort, but possessed no significant or permanent risk of harm. Severe= Interrupted activities of daily living significantly affected clinical status or required intensive therapeutic intervention.
Time Frame: DBT Phase: During 12 weeks of treatment
Population: DBT safety analysis set included the participants who were enrolled and took >= 1 dose of DB study drug (zavegepant or placebo), i.e., non-missing study drug start date.
Measure: Count of Participants; unit: Participants
Groups:
- Zavegepant Pooled (DBT): Participants were randomized to receive Zavegepant 100 mg or 200 mg daily for 12 weeks in DBT phase.
Arm/Group | Zavegepant 100 mg (DBT) | Zavegepant 200 mg (DBT) | Zavegepant Pooled (DBT) | Placebo (DBT) Matched to Zavegepant 100 mg | Placebo (DBT) Matched to Zavegepant 200 mg | Placebo Pooled (DBT)
Number analyzed (Participants) | 173 | 175 | 348 | 86 | 88 | 174
Participants | 20 | 25 | 45 | 13 | 9 | 22

9. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs): DBT Phase
Description: AEs: new untoward medical occurrence or worsening of a pre-existing medical condition in participant or clinical investigation participant administered investigational product that does not necessarily have a causal relationship with treatment. SAE was defined as any event that met any of the following criteria: death; life-threatening; inpatient hospitalization or prolongation of existing hospitalization; persistent or significant disability/incapacity; congenital anomaly/birth defect in the offspring of a participant; other important medical events that may not have resulted in death, be life-threatening, or required hospitalization, based upon appropriate medical judgment, they may have jeopardized the participant and may have required medical or surgical intervention.
Time Frame: DBT Phase: During 12 weeks of treatment
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Zavegepant 100 mg (DBT) | Zavegepant 200 mg (DBT) | Zavegepant Pooled (DBT) | Placebo (DBT) Matched to Zavegepant 100 mg | Placebo (DBT) Matched to Zavegepant 200 mg | Placebo Pooled (DBT)
Number analyzed (Participants) | 173 | 175 | 348 | 86 | 88 | 174
Participants | 1 | 1 | 2 | 0 | 1 | 1

10. Secondary Outcome: Number of Participants With AEs Leading to Study Drug Discontinuation: DBT Phase
Description: An AE was defined as any new untoward medical occurrence or worsening of a pre-existing medical condition in a participant or clinical investigation participant administered an investigational (medicinal) product and that does not necessarily have a causal relationship with this treatment.
Time Frame: DBT Phase: During 12 weeks of treatment
Population: DBT safety analysis set included the participants in the who were enrolled and who took >=1 dose of DB study drug (zavegepant or placebo), i.e., non-missing study drug start date.
Measure: Count of Participants; unit: Participants
Arm/Group | Zavegepant 100 mg (DBT) | Zavegepant 200 mg (DBT) | Zavegepant Pooled (DBT) | Placebo (DBT) Matched to Zavegepant 100 mg | Placebo (DBT) Matched to Zavegepant 200 mg | Placebo Pooled (DBT)
Number analyzed (Participants) | 173 | 175 | 348 | 86 | 88 | 174
Participants | 2 | 5 | 7 | 3 | 4 | 7

11. Secondary Outcome: Number of Participants With Grade 3 to 4 Laboratory Test Abnormalities: DBT Phase
Description: Laboratory tests included eosinophils, hemoglobin, leukocytes, lymphocytes, neutrophils, platelets; albumin, alkaline phosphatase, alanine aminotransferase (ALT), aspartate aminotransferase (AST), bicarbonate, bilirubin, calcium, cholesterol, potassium, sodium, triglycerides, uric acid, urinalysis, urine protein, creatine kinase (CK), creatinine, glomerular filtration rate (GFR), glucose, glucose fasting, lactate dehydrogenase, low density lipoprotein (LDL) Cholesterol, LDL Cholesterol. Number of participants with grade 3 to 4 laboratory test abnormalities were evaluated in this outcome measure. Only rows which included at least 1 participant in any reporting group with grade 3 to 4 abnormality were reported in this outcome measure. As per Common Terminology Criteria for Adverse Events (CTCAE version 5.0) Grade 3= severe and Grade 4= life-threatening or disabling.
Time Frame: DBT: During 12 weeks of treatment
Population: DBT safety analysis set included the participants in the who were enrolled and who took >=1 dose of DB study drug (zavegepant or placebo), i.e., non-missing study drug start date. Participants reported under "Overall Number of Participants Analyzed" contributed data but may not be evaluable for every row and "Number Analyzed" signifies participants evaluable for the specified rows.
Measure: Count of Participants; unit: Participants
Arm/Group | Zavegepant 100 mg (DBT) | Zavegepant 200 mg (DBT) | Zavegepant Pooled (DBT) | Placebo (DBT) Matched to Zavegepant 100 mg | Placebo (DBT) Matched to Zavegepant 200 mg | Placebo Pooled (DBT)
Number analyzed (Participants) | 173 | 175 | 348 | 86 | 88 | 174
Participants
  Hemoglobin: number analyzed (Participants) | 166 | 160 | 326 | 81 | 83 | 164
  Hemoglobin | 0 | 1 | 1 | 0 | 0 | 0
  Creatine Kinase: number analyzed (Participants) | 170 | 168 | 338 | 85 | 85 | 170
  Creatine Kinase | 5 | 7 | 12 | 1 | 0 | 1
  LDL Cholesterol: number analyzed (Participants) | 150 | 147 | 297 | 69 | 73 | 142
  LDL Cholesterol | 7 | 6 | 13 | 2 | 5 | 7
  LDL Cholesterol, fasting: number analyzed (Participants) | 72 | 63 | 135 | 30 | 38 | 68
  LDL Cholesterol, fasting | 4 | 1 | 5 | 1 | 3 | 4
  LDL Cholesterol, not fasting: number analyzed (Participants) | 45 | 49 | 94 | 22 | 21 | 43
  LDL Cholesterol, not fasting | 0 | 3 | 3 | 0 | 1 | 1
  Potassium, high: number analyzed (Participants) | 167 | 161 | 328 | 81 | 83 | 164
  Potassium, high | 0 | 0 | 0 | 3 | 0 | 3
  Triglycerides: number analyzed (Participants) | 150 | 147 | 297 | 69 | 73 | 142
  Triglycerides | 1 | 0 | 1 | 0 | 0 | 0
  Urinalysis: number analyzed (Participants) | 148 | 142 | 290 | 69 | 71 | 140
  Urinalysis | 1 | 0 | 1 | 0 | 0 | 0

12. Secondary Outcome: Number of Participants With Moderate or Severe AEs: OLE Phase
Description: as for outcome 8
Time Frame: OLE: During 52 weeks of treatment
Population: OL safety analysis set included the participants who took >= 1 dose of OL zavegepant, i.e., nonmissing OL zavegepant start date.
Measure: Count of Participants; unit: Participants
Groups:
- Zavegepant 100 mg (OLE): Participants who received Zavegepant 100 mg orally as soft gelatin capsules (25 mg *4 capsules) daily for 52 weeks in OLE phase.
- Zavegepant 200 mg (OLE): Participants who received Zavegepant 200 mg orally as soft gelatin capsules (25 mg *8 capsules) daily for 52 weeks in OLE phase.
Arm/Group | Zavegepant 100 mg (OLE) | Zavegepant 200 mg (OLE)
Number analyzed (Participants) | 155 | 143
Participants | 29 | 37

13. Secondary Outcome: Number of Participants With SAEs: OLE Phase
Description: as for outcome 9
Time Frame: OLE: During 52 weeks of treatment
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Zavegepant 100 mg (OLE) | Zavegepant 200 mg (OLE)
Number analyzed (Participants) | 155 | 143
Participants | 1 | 3

14. Secondary Outcome: Number of Participants With AEs Leading to Study Drug Discontinuation: OLE Phase
Description: as for outcome 10
Time Frame: OLE: During 52 weeks of treatment
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Zavegepant 100 mg (OLE) | Zavegepant 200 mg (OLE)
Number analyzed (Participants) | 155 | 143
Participants | 2 | 4

15. Secondary Outcome: Number of Participants With Grade 3 to 4 Laboratory Test Abnormalities: OLE Phase
Description: as for outcome 11
Time Frame: OLE: During 52 weeks of treatment
Population: OL safety analysis set included the participants who took >= 1 dose of OL zavegepant, i.e., nonmissing OL zavegepant start date. Here, "Number Analyzed" signifies participants evaluable for the specified rows. "Overall Number of Participants Analyzed" contributed data to table but may not have evaluable data for every row.
Measure: Count of Participants; unit: Participants
Arm/Group | Zavegepant 100 mg (OLE) | Zavegepant 200 mg (OLE)
Number analyzed (Participants) | 155 | 143
Participants
  Hemoglobin: number analyzed (Participants) | 149 | 136
  Hemoglobin | 0 | 1
  Neutrophils: number analyzed (Participants) | 149 | 136
  Neutrophils | 1 | 1
  AST: number analyzed (Participants) | 152 | 139
  AST | 0 | 1
  Creatine Kinase: number analyzed (Participants) | 152 | 139
  Creatine Kinase | 10 | 7
  Glucose fasting, low: number analyzed (Participants) | 87 | 78
  Glucose fasting, low | 1 | 0
  LDL Cholesterol: number analyzed (Participants) | 109 | 107
  LDL Cholesterol | 7 | 8
  LDL Cholesterol, fasting: number analyzed (Participants) | 48 | 53
  LDL Cholesterol, fasting | 4 | 4
  LDL Cholesterol, not fasting: number analyzed (Participants) | 32 | 25
  LDL Cholesterol, not fasting | 1 | 1
  Potassium, high: number analyzed (Participants) | 149 | 134
  Potassium, high | 0 | 2
  Triglycerides: number analyzed (Participants) | 109 | 107
  Triglycerides | 1 | 1
  Triglycerides, fasting: number analyzed (Participants) | 48 | 53
  Triglycerides, fasting | 0 | 1
  Triglycerides, not fasting: number analyzed (Participants) | 32 | 25
  Triglycerides, not fasting | 1 | 0
  Urinalysis: number analyzed (Participants) | 108 | 101
  Urinalysis | 1 | 0

16. Secondary Outcome: Percentage of Participants With AST or ALT Elevations >3 * ULN With Total Bilirubin > 2 * ULN: DBT Phase
Description: Elevations of AST or alanine aminotransferase (ALT) > 3 *upper limit of normal (ULN) concurrent with total bilirubin (TBL) > 2 *ULN (elevations on the same laboratory collection date) were included.
Time Frame: DBT: Over 12 weeks of treatment
Population: as for outcome 10
Measure: Number (97.5% Confidence Interval); unit: Percentage of participants
Arm/Group | Zavegepant 100 mg (DBT) | Zavegepant 200 mg (DBT) | Zavegepant Pooled (DBT) | Placebo (DBT) Matched to Zavegepant 100 mg | Placebo (DBT) Matched to Zavegepant 200 mg | Placebo Pooled (DBT)
Number analyzed (Participants) | 173 | 175 | 348 | 86 | 88 | 174
Percentage of participants | 0 [0.0 to 2.5] | 0 [0.0 to 2.5] | 0 [0.0 to 1.3] | 0 [0.0 to 5.0] | 0 [0.0 to 4.9] | 0 [0.0 to 2.5]

17. Secondary Outcome: Percentage of Participants With AST or ALT Elevations >3 * ULN With Total Bilirubin > 2 * ULN: OLE Phase
Description: Elevations of AST or ALT > 3 * ULN concurrent with TBL > 2 *ULN were defined as elevations on the same collection date.
Time Frame: OLE: Over 52 weeks of treatment
Population: as for outcome 12
Measure: Number (97.5% Confidence Interval); unit: Percentage of participants
Arm/Group | Zavegepant 100 mg (OLE) | Zavegepant 200 mg (OLE)
Number analyzed (Participants) | 155 | 143
Percentage of participants | 0 [0.0 to 2.8] | 0 [0.0 to 3.0]

18. Secondary Outcome: Number of Participants With Hepatic-related AEs by Intensity: DBT Phase
Description: An AE was defined as any new untoward medical occurrence or worsening of a pre-existing medical condition in a participant or clinical investigation participant administered an investigational (medicinal) product and that does not necessarily have a causal relationship with this treatment. AEs by intensity: Mild: Transient and may require only minimal treatment or therapeutic intervention. Event did not interfere with activities of daily living. Moderate: Alleviated with additional specific therapeutic intervention. Event interfered with activities of daily living, causing discomfort, but possessed no significant or permanent risk of harm. Severe: Interrupted activities of daily living significantly affected clinical status or required intensive therapeutic intervention.
Time Frame: DBT Phase: During 12 weeks of treatment
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Zavegepant 100 mg (DBT) | Zavegepant 200 mg (DBT) | Zavegepant Pooled (DBT) | Placebo (DBT) Matched to Zavegepant 100 mg | Placebo (DBT) Matched to Zavegepant 200 mg | Placebo Pooled (DBT)
Number analyzed (Participants) | 173 | 175 | 348 | 86 | 88 | 174
Participants
  Mild | 1 | 0 | 1 | 1 | 0 | 1
  Moderate | 0 | 0 | 0 | 1 | 0 | 1
  Severe | 0 | 0 | 0 | 0 | 0 | 0

19. Secondary Outcome: Number of Participants With Hepatic-related AEs Leading to Study Drug Discontinuation: DBT Phase
Description: as for outcome 10
Time Frame: DBT Phase: During 12 weeks of treatment
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Zavegepant 100 mg (DBT) | Zavegepant 200 mg (DBT) | Zavegepant Pooled (DBT) | Placebo (DBT) Matched to Zavegepant 100 mg | Placebo (DBT) Matched to Zavegepant 200 mg | Placebo Pooled (DBT)
Number analyzed (Participants) | 173 | 175 | 348 | 86 | 88 | 174
Participants | 0 | 0 | 0 | 0 | 0 | 0

20. Secondary Outcome: Number of Participants With Hepatic-related AEs by Intensity: OLE Phase
Description: as for outcome 18
Time Frame: OLE: Over 52 weeks of treatment
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Zavegepant 100 mg (OLE) | Zavegepant 200 mg (OLE)
Number analyzed (Participants) | 155 | 143
Participants
  Mild | 1 | 1
  Moderate | 1 | 2
  Severe | 0 | 1

21. Secondary Outcome: Number of Participants With Hepatic-related AEs Leading to Study Drug Discontinuation: OLE Phase
Description: as for outcome 10
Time Frame: OLE: Over 52 weeks of treatment
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Zavegepant 100 mg (OLE) | Zavegepant 200 mg (OLE)
Number analyzed (Participants) | 155 | 143
Participants | 0 | 1

ADVERSE EVENTS:
Time Frame: DBT Phase: 12 weeks of treatment; OLE Phase: 52 weeks of treatment; Follow-up phase: 8 weeks after the discontinuation or completion of treatment in DBT (if not entered OLE) or OLE phase
Groups:
- Zavegepant 100 mg (DBT): Participants were randomized to receive Zavegepant 100 mg orally as soft gelatin capsules (25 mg *4 capsules) daily for 12 weeks in DBT phase.
- Zavegepant 100 mg DBT/Zavegepant 100 mg OLE: Follow-up: Participants who received Zavegepant 100 mg in DBT phase or in DBT and OLE phases and were followed up for safety for 8 weeks post discontinuation or completion of treatment in DBT or OLE phase.
- Zavegepant 200 mg DBT/ Zavegepant 200 mg OLE: Follow-up: Participants who received Zavegepant 200 mg in DBT phase or in DBT and OLE phases and were followed up for safety for 8 weeks post discontinuation or completion of treatment in DBT or OLE phase.
- Placebo Matched to Zavegepant 100 mg (DBT)/ Zavegepant 100 mg OLE: Follow-up: Participants who received Placebo matched to Zavegepant 100 mg in DBT phase or Placebo matched to Zavegepant 100 mg in DBT phase and Zavegepant 100 mg in OLE phase, were followed up for safety for 8 weeks post discontinuation or completion of treatment in DBT or OLE phase.
- Placebo Matched to Zavegepant 200 mg (DBT)/ Zavegepant 200 mg OLE: Follow-up: Participants who received Placebo matched to Zavegepant 200 mg in DBT phase or Placebo matched to Zavegepant 200 mg in DBT phase and Zavegepant 200 mg in OLE phase, were followed up for safety for 8 weeks post discontinuation or completion of treatment in DBT or OLE phase.
- Placebo Pooled (DBT)/No Zavegepant OLE: Follow-up: Participants who received Placebo matched to Zavegepant 100 mg or 200 mg in DBT phase and no Zavegepant in OLE phase were followed up for safety for 8 weeks post discontinuation or completion of treatment in DBT phase.
Arm/Group | Zavegepant 100 mg (DBT) | Zavegepant 200 mg (DBT) | Zavegepant Pooled (DBT) | Placebo (DBT) Matched to Zavegepant 100 mg | Placebo (DBT) Matched to Zavegepant 200 mg | Placebo Pooled (DBT) | Zavegepant 100 mg (OLE) | Zavegepant 200 mg (OLE) | Zavegepant 100 mg DBT/Zavegepant 100 mg OLE: Follow-up | Zavegepant 200 mg DBT/ Zavegepant 200 mg OLE: Follow-up | Placebo Matched to Zavegepant 100 mg (DBT)/ Zavegepant 100 mg OLE: Follow-up | Placebo Matched to Zavegepant 200 mg (DBT)/ Zavegepant 200 mg OLE: Follow-up | Placebo Pooled (DBT)/No Zavegepant OLE: Follow-up
All-Cause Mortality (participants affected / at risk) | 1/173 | 0/175 | 0/348 | 0/86 | 0/88 | 0/174 | 0/155 | 0/143 | 0/154 | 0/162 | 0/47 | 0/48 | 0/70
Serious Adverse Events (participants affected / at risk) | 1/173 | 1/175 | 2/348 | 0/86 | 1/88 | 1/174 | 1/155 | 3/143 | 0/154 | 1/162 | 1/47 | 0/48 | 0/70
Other Adverse Events (participants affected / at risk) | 14/173 | 8/175 | 22/348 | 13/86 | 11/88 | 24/174 | 12/155 | 12/143 | 0/154 | 0/162 | 0/47 | 0/48 | 0/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Zavegepant 100 mg (DBT) (N=173) | Zavegepant 200 mg (DBT) (N=175) | Zavegepant Pooled (DBT) (N=348) | Placebo (DBT) Matched to Zavegepant 100 mg (N=86) | Placebo (DBT) Matched to Zavegepant 200 mg (N=88) | Placebo Pooled (DBT) (N=174) | Zavegepant 100 mg (OLE) (N=155) | Zavegepant 200 mg (OLE) (N=143) | Zavegepant 100 mg DBT/Zavegepant 100 mg OLE: Follow-up (N=154) | Zavegepant 200 mg DBT/ Zavegepant 200 mg OLE: Follow-up (N=162) | Placebo Matched to Zavegepant 100 mg (DBT)/ Zavegepant 100 mg OLE: Follow-up (N=47) | Placebo Matched to Zavegepant 200 mg (DBT)/ Zavegepant 200 mg OLE: Follow-up (N=48) | Placebo Pooled (DBT)/No Zavegepant OLE: Follow-up (N=70)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertensive heart disease (Cardiac disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Zavegepant 100 mg (DBT) (N=173) | Zavegepant 200 mg (DBT) (N=175) | Zavegepant Pooled (DBT) (N=348) | Placebo (DBT) Matched to Zavegepant 100 mg (N=86) | Placebo (DBT) Matched to Zavegepant 200 mg (N=88) | Placebo Pooled (DBT) (N=174) | Zavegepant 100 mg (OLE) (N=155) | Zavegepant 200 mg (OLE) (N=143) | Zavegepant 100 mg DBT/Zavegepant 100 mg OLE: Follow-up (N=154) | Zavegepant 200 mg DBT/ Zavegepant 200 mg OLE: Follow-up (N=162) | Placebo Matched to Zavegepant 100 mg (DBT)/ Zavegepant 100 mg OLE: Follow-up (N=47) | Placebo Matched to Zavegepant 200 mg (DBT)/ Zavegepant 200 mg OLE: Follow-up (N=48) | Placebo Pooled (DBT)/No Zavegepant OLE: Follow-up (N=70)
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 3 | 1 | 5 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 12 | 5 | 17 | 8 | 5 | 13 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 2 | 1 | 3 | 6 | 1 | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 12 | 12 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2022-05-16): https://cdn.clinicaltrials.gov/large-docs/33/NCT04804033/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-30): https://cdn.clinicaltrials.gov/large-docs/33/NCT04804033/SAP_001.pdf